CLINICAL TRIAL: NCT06256588
Title: A Randomized, Double-blind, Placebo-controlled Phase 3 Study to Evaluate Dostarlimab as Sequential Therapy After Chemoradiation in Participants With Locally Advanced Unresected Head and Neck Squamous Cell Carcinoma
Brief Title: A Study of Dostarlimab vs Placebo After Chemoradiation in Adult Participants With Locally Advanced Unresected Head and Neck Squamous Cell Carcinoma
Acronym: JADE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 221530; 2023-508613-17 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Neoplasms, Head and Neck
Keywords: JEMPERLI; Dostarlimab; Placebo; Chemoradiation; HNSCC
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — dostarlimab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Dostarlimab (Experimental)
  Interventions: Drug: Dostarlimab
- Arm B: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dostarlimab — Dostarlimab will be administered as an intravenous (IV) infusion
  Arms: Arm A: Dostarlimab
Drug: Placebo — Placebo will be administered as an IV infusion
  Arms: Arm B: Placebo

SUMMARY:
The goal of this study is to assess the safety and effectiveness of Dostarlimab compared to Placebo in adult participants with Head and Neck Squamous Cell Carcinoma (HNSCC)

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

* Has newly diagnosed unresected Locally Advanced (LA) histologically confirmed HNSCC of the oral cavity, oropharynx, hypopharynx or larynx and completed cisplatin plus radiotherapy (termed "CRT" in this protocol) with curative intent and has no evidence of distant metastatic disease.
* Has provided acceptable core or excisional biopsy obtained prior to CRT:

  * PD-L1 positive tumor status
  * If the primary tumor site is oropharyngeal carcinoma, the participant must have p16 immunohistochemistry (IHC) testing.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Has adequate organ function.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Has received prior radiation therapy (RT), systemic therapy, targeted therapy, or surgery for management of head and neck cancer not considered part of CRT. Participants receiving induction chemotherapy are excluded. CRT combinations with components other than cisplatin and RT (e.g., experimental agents, including radiosensitizers/radioprotectants, cetuximab) are not eligible.
* Has cancer outside of the oropharynx, larynx, hypopharynx or oral cavity, such as nasopharyngeal, sinus, other para-nasal, or other unknown primary head and neck cancer. Has more than one primary HNSCC tumor.
* Has experienced any of the following with prior immunotherapy: any immune-related adverse event (irAE) of Grade ≥3, immune-related severe neurologic events of any grade (e.g., myasthenic syndrome/myasthenia gravis, encephalitis, Guillain-Barré Syndrome, or transverse myelitis), exfoliative dermatitis of any grade (Stevens-Johnson Syndrome, toxic epidermal necrolysis, or Drug Rash with Eosinophilia and Systemic Symptoms [DRESS] syndrome), or myocarditis of any grade. Non-clinically significant laboratory abnormalities are not exclusionary.
* Has undergone any major surgical procedure or experienced significant traumatic injury that has not resolved by the time of randomization.
* Has any history of interstitial lung disease or pneumonitis (past or current).
* Has cirrhosis of any stage or current unstable liver biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal/gastric varices, or persistent jaundice.
* Has a history or current evidence of any medical condition, therapy, or laboratory abnormality that might confound the study results, interfere with their participation for the full duration of the study intervention, or indicate it is not in the best interest of the participant to participate, in the opinion of the investigator.
* Is receiving any other anticancer or experimental therapy. No other experimental therapies (including but not limited to chemotherapy, radiation, hormonal treatment, antibody therapy, immunotherapy, gene therapy, vaccine therapy, or other experimental drugs) of any kind are permitted while the participant is receiving study intervention.
* Previous treatment with anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or an agent directed to another stimulatory or coinhibitory T-cell receptor [e.g., Cytotoxic T-lymphocyte associated protein 4 (CTLA4), OX-40, CD137]
* Is pregnant, breastfeeding, or expecting to conceive children within the projected duration of the study, starting with the Screening Visit through 120 days after the last dose of study intervention.
* Has a history of severe allergic and/or anaphylactic reactions to chimeric, human or humanized antibodies, fusion proteins, or known allergies to dostarlimab or its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 864 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2029-10-26 (Estimated)

PRIMARY OUTCOMES:
Event-free Survival (EFS) Assessed by Blinded Independent Central Review (BICR) | Up to approximately 5 years
  Event Free Survival (EFS) is defined as the time from the date of randomization to the date of an event, where an event is defined as locoregional progression or recurrence, or distant metastasis per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as per BICR; Salvage surgery at the primary tumor site; Neck dissection or surgery performed >20 weeks after completion of Concomitant Chemoradiotherapy (CRT) when invasive cancer is present or Death from any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 5 years
  OS is defined as the time from date of randomization to the date of death by any cause.
Event-free Survival (EFS) assessed by investigator | Up to approximately 5 years
  Event Free Survival (EFS) is defined as the time from the date of randomization to the date of an event as per primary endpoint, however with investigator assessment per RECIST 1.1
Number of Participants with treatment emergent adverse events (TEAEs), Immune-mediated TEAEs, and serious adverse events (SAEs) by severity | Up to approximately 5 years
Number of Participants with TEAEs and SAEs leading to dose delays, withdrawals or death | Up to approximately 5 years
Number of participants with clinically significant changes in laboratory, vital signs, and safety assessment parameters | Up to approximately 5 years
Serum Concentration of Dostarlimab | Up to approximately 15 months
Serum Concentration of Dostarlimab at End of Infusion (C-EoI) | Up to approximately 15 months
Serum Predose trough concentration (Ctrough) of Dostarlimab | Up to approximately 15 months
Number of Participants with Anti-Drug Antibodies against Dostarlimab | Up to approximately 15 months

CONTACTS AND LOCATIONS:
Locations (208):
- United States (29):
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Solvang, California
  - GSK Investigational Site, Stockton, California
  - GSK Investigational Site, Torrance, California
  - GSK Investigational Site, Farmington, Connecticut
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Tamarac, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Fort Wayne, Indiana
  - GSK Investigational Site, Iowa City, Iowa
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Germantown, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Fredericksburg, Virginia
  - GSK Investigational Site, Wytheville, Virginia
  - GSK Investigational Site, Tacoma, Washington
- Argentina (7):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aire
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Rosario
  - GSK Investigational Site, San Juan
  - GSK Investigational Site, San Miguel de Tucumán
  - GSK Investigational Site, Viedma
- Australia (6):
  - GSK Investigational Site, Blacktown, New South Wales
  - GSK Investigational Site, Douglas, Queensland
  - GSK Investigational Site, Herston, Queensland
  - GSK Investigational Site, Ballarat, Victoria
  - GSK Investigational Site, Geelong, Victoria
  - GSK Investigational Site, Melbourne, Victoria
- Belgium (5):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Charleroi
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Yvoir
- Brazil (12):
  - GSK Investigational Site, Barretos
  - GSK Investigational Site, Belo Horizonte
  - GSK Investigational Site, Florianópolis
  - GSK Investigational Site, Ijuí
  - GSK Investigational Site, Jaú
  - GSK Investigational Site, Joinville
  - GSK Investigational Site, Natal
  - GSK Investigational Site, Porto Alegre
  - GSK Investigational Site, Salvador
  - GSK Investigational Site, São José do Rio Preto
  - GSK Investigational Site, São Paulo
  - GSK Investigational Site, Vitória
- Canada (3):
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- China (21):
  - GSK Investigational Site, Chongqing, Chongqing Municipality
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Changsha
  - GSK Investigational Site, Changzhou
  - GSK Investigational Site, Chengdu
  - GSK Investigational Site, Dongguan
  - GSK Investigational Site, Fuzhou
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Hefei
  - GSK Investigational Site, Hengyang
  - GSK Investigational Site, Jinan
  - GSK Investigational Site, Linyi
  - GSK Investigational Site, Nanchang
  - GSK Investigational Site, Nanning
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Taiyuan
  - GSK Investigational Site, Wuhan
  - GSK Investigational Site, Xiamen
  - GSK Investigational Site, Zhengzhou
  - GSK Investigational Site, Zhuhai
- Czechia (3):
  - GSK Investigational Site, Olomouc
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Zlín
- France (8):
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Poitiers
  - GSK Investigational Site, Quimper
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Rouen
  - GSK Investigational Site, Vandœuvre-lès-Nancy
- Germany (8):
  - GSK Investigational Site, Augsburg
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Erlangen
  - GSK Investigational Site, Essen
  - GSK Investigational Site, Giessen
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Neuruppin
  - GSK Investigational Site, Straubing
- Greece (3):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Larissa
  - GSK Investigational Site, Thessaloniki
- Hungary (3):
  - GSK Investigational Site, Győr
  - GSK Investigational Site, Kaposvár
  - GSK Investigational Site, Nyíregyháza
- India (8):
  - GSK Investigational Site, Bengaluru
  - GSK Investigational Site, Bhubaneswar
  - GSK Investigational Site, Hyderabad
  - GSK Investigational Site, Mumbai
  - GSK Investigational Site, Nashik
  - GSK Investigational Site, Nehru Nagar Belagavi Karnataka 590010
  - GSK Investigational Site, Surat
  - GSK Investigational Site, Vijayawada
- Israel (4):
  - GSK Investigational Site, Ashdod
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Jerusalem
  - GSK Investigational Site, Tel Aviv
- Italy (8):
  - GSK Investigational Site, Bologna
  - GSK Investigational Site, Milan
  - GSK Investigational Site, Napoli
  - GSK Investigational Site, Pavia
  - GSK Investigational Site, Prato
  - GSK Investigational Site, Roma
  - GSK Investigational Site, Rozzano MI
  - GSK Investigational Site, Savona
- Japan (19):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Aomori
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kyoto
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Niigata
  - GSK Investigational Site, Numakunai
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Tottori
- Mexico (3):
  - GSK Investigational Site, Guadalajara
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, Oaxaca City
- Norway (3):
  - GSK Investigational Site, Bergen
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Troms
- Poland (7):
  - GSK Investigational Site, Bielsko-Biala
  - GSK Investigational Site, Gliwice
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Przemyśl
  - GSK Investigational Site, Siedlce
  - GSK Investigational Site, Warsaw
- Portugal (6):
  - GSK Investigational Site, Coimbra
  - GSK Investigational Site, Faro
  - GSK Investigational Site, Lisbon
  - GSK Investigational Site, Matosinhos Municipality
  - GSK Investigational Site, Porto
  - GSK Investigational Site, Vila Nova de Gaia
- Romania (8):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Floreşti
  - GSK Investigational Site, Iași
  - GSK Investigational Site, Oradea
  - GSK Investigational Site, Piteşti
  - GSK Investigational Site, Suceava
  - GSK Investigational Site, Timișoara
- South Korea (4):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon Gyeonggi-do
- Spain (12):
  - GSK Investigational Site, BaracaldoVizcaya
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Cartagena Murcia
  - GSK Investigational Site, HebrOn
  - GSK Investigational Site, Jerez de la Frontera
  - GSK Investigational Site, L'Hospitalet de Llobrega
  - GSK Investigational Site, Lugo
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Pamplona
  - GSK Investigational Site, Salamanca
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Zaragoza
- Sweden (3):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Stockholm
  - GSK Investigational Site, Uppsala
- Taiwan (4):
  - GSK Investigational Site, Changhua
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
- Turkey (Türkiye) (5):
  - GSK Investigational Site, Adapazarı
  - GSK Investigational Site, Ankara
  - GSK Investigational Site, Antalya
  - GSK Investigational Site, Istanbul
  - GSK Investigational Site, Istanbul, Şişli
- United Kingdom (6):
  - GSK Investigational Site, Edinburgh
  - GSK Investigational Site, Gloucester
  - GSK Investigational Site, London
  - GSK Investigational Site, Nottingham
  - GSK Investigational Site, Sutton
  - GSK Investigational Site, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/

REFERENCES:
- [Derived] Siu LL, Burtness B, Harrington K, Psyrri A, Saba NF, Tahara M, Carlson G, Dhar A, Grimshaw M, Hua L, Iadevaia R, Theti D, Vlahovic G, Machiels JP. JADE: phase 3 study of sequential dostarlimab post chemoradiotherapy in patients with locally advanced unresected HNSCC. Future Oncol. 2026 Jan 30:1-8. doi: 10.1080/14796694.2026.2619653. Online ahead of print. PMID 41612885